CLINICAL TRIAL: NCT00897351
Title: Evaluation of Polymorphisms, Mutations, and Protein Expression by Automated Quantitative Immunohistochemistry (AQUA) in the LapatinibTargets and Metabolic Pathway in Samples From E5803
Brief Title: Study of Tissue and Blood Samples From Patients With Recurrent Prostate Cancer Who Received Lapatinib on Clinical Trial ECOG-E5803
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000600985; ECOG-E5803T1
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Amplified Fragment Length Polymorphism Analysis; Immunohistochemistry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: mutation analysis
Genetic: polymorphism analysis
Genetic: protein expression analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue and blood in the laboratory from patients with cancer may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research study is looking at tissue and blood samples from patients with recurrent prostate cancer who received lapatinib on clinical trial ECOG-E5803.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the association between polymorphisms in drug metabolizing enzymes and lapatinib ditosylate-associated toxicity in patients with hormone-sensitive recurrent prostate cancer receiving lapatinib ditosylate on clinical trial ECOG-E5803.
* To determine the association between mutations in EGFR, HER-2 and Kras; protein expression of HER2, EGFR, MAPK and AKT; polymorphism controlling androgen synthesis; and progression-free survival.

OUTLINE: Tissue and blood samples collected from patients enrolled on clinical trial ECOG-E5803 are analyzed for correlative studies. Samples are assessed for HER2, EGFR, MAPK, and Akt; EGFR mutations and polymorphisms in CYP3A4; Ras mutations; recently identified mutations in HER2-neu and Kras; and additional polymorphisms in the lapatinib ditosylate metabolic pathway by automated quantitative IHC. Predictors of efficacy and toxicity are analyzed, including markers in the EGFR pathway as predictors of progression-free survival.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of prostate cancer

  * Recurrent disease
* Received lapatinib ditosylate on clinical trial ECOG-E5803

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples submitted for research from patients enrolled on E5803
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2008-07-10 (Actual); Primary Completion 2009-02-10 (Actual); Study Completion 2009-02-10 (Actual)

PRIMARY OUTCOMES:
Polymorphisms associated with toxicity | 1 month
Association between mutations in EGFR, HER-2 and Kras; protein expression of HER2, EGFR, MAPK and AKT; polymorphism controlling androgen synthesis; and progression-free survival | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Jill Kolesar, PharmD, Study Chair — University of Wisconsin, Madison